CLINICAL TRIAL: NCT07124988
Title: Results of Different Modalities of Palatomaxillary Reconstruction , Prospective Comparative Study
Brief Title: Results of Different Modalities of Palatomaxillary Reconstruction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdallah Abozaid, Assistant lecturer of otorhinolaryngology at sohag university hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh_Med_25_7_1MD
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Cancer Maxilla

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- regional flap group 1 (Active Comparator): Regional flap for palatomaxillary defects as Temporalis muscle
  Interventions: Procedure: regional flap
- Distant flap group 2 (Active Comparator): Distant flap for palatomaxillary defects as Radial forearm free flap
  Interventions: Procedure: distant flap

INTERVENTIONS:
Procedure: regional flap — regional flap reconstruction for palatomaxillary defects
  Arms: regional flap group 1
Procedure: distant flap — Distant flap reconstruction for palatomaxillary defects
  Arms: Distant flap group 2

SUMMARY:
Results of different modalities of reconstruction after maxillectomy , prospective comparative study

ELIGIBILITY:
Inclusion Criteria:

* all patients who will undergo maxillectomy (either limited, subtotal or total) due to cancer maxilla ,benign lesions with aggressive behavior ,osteomyelitis, cancer in the surrounding tissues or palatomaxillary trauma.

Exclusion Criteria:maxillary defects of congenital causes

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2027-02-27 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
Mouth opening | 6 months post operative
  measures maximal inter incisional distance to :
  1. normal (more than 35 mm)
  2. mild restriction (20 to 35mm)
  3. moderate restriction (10 to 20 mm)
  4. severe restriction (less than 10 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelkader, professor, Study Chair — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 18 monthes